CLINICAL TRIAL: NCT04849975
Title: Comparison of Pelvimetric Measurements Between MRI and Low-dose Stereoradiography (EOS® Imaging System)
Acronym: CAPEOS®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC21.001
Record Dates: First submitted 2021-03-11; First posted 2021-04-20 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Breech Fetal Presentation
Keywords: Breech Fetal Presentation; MRI; EOS imaging system; Pelvimetric measurements
MeSH Terms: conditions — Breech Presentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pelvimetry group (Experimental): The participants oh this group will successively perform MRI pelvimetry and EOS imaging.
  Interventions: Other: Pelvimetric measurements

INTERVENTIONS:
Other: Pelvimetric measurements — The patients in this group are pregnant women after failure of external manual version (EMV) in case of breech fetal presentation. The participants will successively perform MRI pelvimetry (conventional management) and EOS imaging.

SUMMARY:
The main objective of this study is to compare pelvimetric measurements performed by Magnetic Resonance Imaging (MRI) and by the EOS imaging system.

DETAILED DESCRIPTION:
During pregnancy, after failure of External Manual Version (EMV) in case of breech fetal presentation, a radiological pelvimetry is performed to evaluate the measurements of the pelvis and decide on the appropriate mode of delivery.

Several imaging modalities are used, including pelvic computed tomography (CT),and magnetic resonance imaging (MRI) of the pelvis.

CT scan has the disadvantage of maternal irradiation and MRI has the disadvantage of an inaccurate morphological analysis.The EOS® system is an imaging tool used in radiopediatric to allow precise morphological analysis of bone masses with minimal irradiation.

The quality of the morphological analysis and measurements provided by the EOS® imaging system is the reason for proposing this study comparing the pelvimetric measurements obtained by MRI and by the EOS® imaging system.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Patient requiring pelvimetry (breech fetus)
* Gestation > 36 SA (weeks of amenorrhea)
* Patients with BMI < 35
* Affiliated to social security or similarly regime
* Patients who gave their consent to participate in the study (Patient having agreed to perform both examinations: MRI and EOS system)

Exclusion Criteria:

* Patient with a contraindication to MRI (claustrophobia, pace-maker, intracorporeal metallic element)
* Patient with a contraindication to performing EOS® (person not standing alone)
* Patient who are in exlusion period of another interventiionnal study
* Person deprived of freedom by judicial or administrative decision; person hospitalized for psychitric care; person under legal protection measure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Estimation of the reliability of pelvimetric measurements using Transverse Inlet Diameter measurement | Up to 1 day
  Transverse Inlet Diameter Measurement obtained by EOS® system versus MRI is evaluated in millimeters.
Estimation of the reliability of pelvimetric measurements using ante posterior diameter measurement | Up to 1 day
  Ante posterior diameter of the pelvic inlet obtained by using EOS® system versus MRI is evaluated in millimeters.
Estimation of the reliability of pelvimetric measurements using BiSpinous Diameter measurement | Up to 1 day
  BiSpinous Diameter obtained by EOS® system versus MRI is evaluated in millimeters.
Estimation of the reliability of pelvimetric measurements using Bi-ischiatic mesurement | Up to 1 day
  Bi-ischiatic measurement obtained by EOS® system versus MRI is evaluated in millimeters.
Estimation of the reliability of pelvimetric measurements using Magin's Index calculation | Up to 1 day
  Magnin's Index calculation obtained by using EOS® system versus MRI is evaluated in millimeters.

SECONDARY OUTCOMES:
Pelvis morphological description using Cadwell and Moloy classification | Up to 1 day
  Caldwell and Moloy classification (scale) obtained by MRI and EOS® system is qualified.
Pelvis morphological description using subpubic angle measurement | Up to 1 day
  The measurement of the subpubic angle (in degree) obtained by MRI and EOS® system is qualified.
Pelvis morphological description using obturating holes appearance | Up to 1 day
  The appearance of the obturating holes (descriptive analysis) obtained by MRI and EOS® system is qualified.
Characterization of radiation doses received by EOS® system. | Up to 1 day
  Estimation of irradiation
Evaluation of the intra and inter-observer reproducibility for radiological interpretation | 4 days
  Blind independent reading of MRI and EOS® images by two radiologists on two different days.
Evaluation of the intra and inter-observer reproducibility for clinical interpretation | 4 days
  Blind independent reading of MRI and EOS® images by two independent clinician on two different days with conclusion on the mode of delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Didier R RIETHMULLER, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Pr Riethmuller Didier, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aubry S, Padoin P, Petegnief Y, Vidal C, Riethmuller D, Delabrousse E. Can three-dimensional pelvimetry using low-dose stereoradiography replace low-dose CT pelvimetry? Diagn Interv Imaging. 2018 Sep;99(9):569-576. doi: 10.1016/j.diii.2018.02.008. Epub 2018 Mar 19. PMID 29567122